CLINICAL TRIAL: NCT04702776
Title: Non Inferiority Phase IV Clinical Study, to Compare the Efficacy of the Ophthalmic Solution Humylub Ofteno® PF Against Hyabak® and Lagricel Ofteno® PF When Applied on the Ocular Surface of Patients With Mild to Moderate Dry Eye.
Brief Title: Study to Compare the Efficacy of the Ophthalmic Solution Humylub Ofteno® PF With Hyabak® and Lagricel Ofteno® PF as Treatment for Dry Eye.
Acronym: PRO-087
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH087-0120/IV
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Phase IV, non inferiority, controlled, open, comparative, multicenter clinical study
Who Masked: Participant, Investigator
Masking Description: After signing the informed consent form (ICF), every subject will receive a coded patient number and will be assigned randomly to one of the investigation products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1; Humylub Ofteno® PF (Experimental): Humylub Ofteno® PF (sodium hyaluronate 0.1%/chondroitin sulfate 0.18%) ophthalmic solution applied QID for 30 days.
  Interventions: Drug: Sodium hyaluronate 0.1%/chondroitin sulfate 0.18%
- Arm 2; Hyabak® (Active Comparator): Hyabak® PF (sodium hyaluronate 0.15%) ophthalmic solution applied QID for 30 days.
  Interventions: Drug: Sodium hyaluronate 0.15%
- Arm 3; Lagricel Ofteno® PF (Active Comparator): Lagricel Ofteno® PF (sodium hyaluronate 0.4%) ophthalmic solution applied QID for 30 days.
  Interventions: Drug: Sodium hyaluronate 0.4%

INTERVENTIONS:
Drug: Sodium hyaluronate 0.1%/chondroitin sulfate 0.18% — Application of one drop of Humylub Ofteno® PF (Sodium hyaluronate 0.1%/chondroitin sulfate 0.18%) QID in both eyes (OU) during 30 days.
  Other Names: Humylub Ofteno® PF; PRO-087
  Arms: Arm 1; Humylub Ofteno® PF
Drug: Sodium hyaluronate 0.15% — Application of one drop of Hyabak® PF (Sodium hyaluronate 0.15%) QID in OU during 30 days.
  Other Names: Hyabak® PF
  Arms: Arm 2; Hyabak®
Drug: Sodium hyaluronate 0.4% — Application of one drop of Lagricel Ofteno® PF (Sodium Hyaluronate 0.4%) QID in OU during 30 days.
  Other Names: Lagricel Ofteno® PF; PRO-037
  Arms: Arm 3; Lagricel Ofteno® PF

SUMMARY:
Phase IV, non inferiority, controlled, open, multicenter clinical study to compare the efficacy of the Ophthalmic Solution Humylub Ofteno® PF against Hyabak® and Lagricel Ofteno® PF applied quater in die (QID) for 30 days in patients with mild to moderate dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Age ≥ 18 years old
* Women in child-bearing age must assure the continuation (start ≥ 30 days prior to informed consent signing) of a hormonal contraceptive method or intrauterine device (IUD) during the study.
* Presenting a mild to moderate dry eye disease diagnosis, defined as:

  * OSDI score ≥ 13, plus one of the following:

    * More than 5 dots of corneal staining
    * More than 9 dots of conjunctival staining
    * Tear break-up time < 10 seconds

Exclusion Criteria:

* - Pregnancy, breastfeeding or planning to become pregnant during the time of the study
* Having participated in clinical trials within 30 days prior to the eligibility visit.
* Having participated previously in this study.
* BCVA equal or worse than 20/200, in either eye.
* Diagnosis of any of the following:

  * Allergic, viral or bacterial conjunctivitis
  * Anterior blepharitis
  * Parasite infestation of any ocular or annex structures (Demodex, for example)
  * Unresolved history of ocular trauma
  * Scarring diseases of the ocular surface
  * Corneal or conjunctival ulcers
  * Filamentary keratitis
  * Neurotrophic keratitis
  * Bullous keratopathy
  * Neoplastic diseases of the ocular surface or ocular annexes
  * Diseases presenting fibrovascular proliferations on the corneal or conjunctival surface.
  * Any retinal or posterior segment diseases that require treatment or threat the visual outcome.
  * Glaucoma
  * Any palpebral alteration that causes eyelid malposition, limiting the adequate closure or aperture of this structures, or that cause tearing.
* Requiring management for dry eye that includes implementation of treatments described in the step 2 management recommendations of the Tear Film & Ocular Surface Society's Dry Eye Work Shop II (TFO DEWS II).
* Previous history of drug addiction within the last 2 years prior to signing this study's informed consent form.
* Having a previous history of any ophthalmological surgical procedure, within the last 3 months prior to the informed consent signing date.
* Being a contact lens user, rigid or soft. Inclusion is possible if the use of contact lenses is suspended both during the study period and at least 15 days prior inclusion takes place.
* Previous history of any medical affliction, acute or chronic, that according to the investigator may increase either the risk to the patient for participating in this study or the risk of interference of the accurate interpretation of results.
* Known hypersensitivity to any of the components of the products used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Clínica de Bioequivalencia, S. de R.L. de C.V., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Garcia-Sanchez G, Jauregui-Franco RO, Quirarte-Justo S, Sanchez-Rios A, Olvera-Montano O. Influence of Environmental Factors with Clinical Signs and Symptoms in the Management of Dry Eye Disease. Clin Ophthalmol. 2024 Aug 30;18:2439-2451. doi: 10.2147/OPTH.S480223. eCollection 2024. PMID 39233999

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The minimun sample size was not reached secondary to follow up loss and protocol deviations. Therefore, the efficacy analysis was performed in an exploratory manner and it was not possible to contrast the hypoteses.
Period: Overall Study
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Started | 61 | 61 | 60
Completed | 56 | 56 | 52
Not Completed | 5 | 5 | 8
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 4
Not completed — Protocol Violation | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF | Total
Number analyzed (Participants) | 61 | 61 | 60 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 61 | 60 | 182
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (11) | 31.7 (11.7) | 31.4 (10.2) | 30.9 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 36 | 102
  Male | 28 | 28 | 24 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Measure Analysis Population Description: Race and Ethnicity were not collected from any participant.
  Participants
    Hispanic or Latino | 61 | 61 | 60 | 182
    Not Hispanic or Latino | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 61 | 61 | 60 | 182
Conjunctival hyperemia [Count of Participants; unit: Participants] | 24 | 19 | 16 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Surface Disease Index (OSDI)
Description: OSDI is a 12-item questionnaire used to evaluate symptoms associated with dry eye disease, as well as classify their severity. According the obtained score, categories are as follows: normal (0-12 points), mild (13-22 points), moderate (23-32 points), or severe (33-100 points). A higher score is a worse outcome. • This outcome measure considered the Per Protocol (PP) population.
Time Frame: Days: 0 (± 2) (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: In total, 18 participants were discontinued from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 46 | 49 | 40
score on a scale
  Elegibility visit | 26.4 (5.1) | 26.3 (5.8) | 26.6 (4.9)
  First follow-up visit | 16.4 (8.3) | 14.0 (10.4) | 15.2 (8.3)
  Final visit | 11.2 (9.4) | 8.8 (7.5) | 10.7 (9.0)

2. Secondary Outcome: Noninvasive Keratograph Break-up Time (NIKBUT)
Description: This evaluation will be performed through an Oculus Keratograph 5M, and the parameter "first break-up time" will be recorded as NIKBUT. A lower value is a worse outcome. This outcome measure considered the Per Protocol (PP) population.
Time Frame: Days: 0 - 2 (baseline visit),17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: In total, 18 participants were discontinued from the study.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 46 | 49 | 40
seconds
  Baseline visit | 6.8 (3.9) | 5.2 (3.0) | 7.1 (4.3)
  First follow-up visit | 7.3 (4.8) | 6.9 (4.8) | 7.7 (4.9)
  Final visit | 8.7 (5.3) | 7.8 (4.9) | 7.1 (3.9)

3. Secondary Outcome: Change of Conjunctival and Corneal Staining With Lissamine Green
Description: The change in proportion of participant's abscence of conjunctival and corneal staining with lissamine green will be analyzed. The evaluation will take place after applying the lissamine green stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V). This outcome measure considered the Per Protocol (PP) population.
Time Frame: Days: 0 (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: In total, 18 participants were discontinued from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 46 | 49 | 40
Participants
  Eligibility visit: 0 | 20 | 23 | 16
  Eligibility visit: I | 21 | 22 | 24
  Eligibility visit: II | 3 | 4 | 0
  Eligibility visit: III | 2 | 0 | 0
  Eligibility visit: IV | 0 | 0 | 0
  First follow-up visit: 0 | 25 | 28 | 25
  First follow-up visit: I | 16 | 19 | 12
  First follow-up visit: II | 4 | 1 | 3
  First follow-up visit: III | 0 | 1 | 0
  First follow-up visit: IV | 1 | 0 | 0
  Final visit: 0 | 33 | 32 | 23
  Final visit: I | 12 | 15 | 17
  Final visit: II | 1 | 2 | 0
  Final visit: III | 0 | 0 | 0
  Final visit: IV | 0 | 0 | 0

4. Secondary Outcome: Change of Conjunctival and Corneal Staining With Fluorescein
Description: The change in proportion of participant's abscence of conjunctival and corneal staining with fluorescein will be analyzed. The evaluation will take place after applying the fluorescein stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V). This outcome measure considered the Per Protocol (PP) population.
Time Frame: Days: 0 (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: In total, 18 participants were discontinued from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 46 | 49 | 40
Participants
  Elegibility visit: 0 | 19 | 20 | 16
  Elegibility visit: I | 19 | 27 | 20
  Elegibility visit: II | 7 | 2 | 4
  Elegibility visit: III | 1 | 0 | 0
  First follow-up visit: 0 | 31 | 23 | 25
  First follow-up visit: I | 12 | 22 | 14
  First follow-up visit: II | 3 | 4 | 1
  First follow-up visit: III | 0 | 0 | 0
  Final visit: 0 | 36 | 34 | 24
  Final visit: I | 10 | 15 | 14
  Final visit: II | 0 | 0 | 2
  Final visit: III | 0 | 0 | 0

5. Secondary Outcome: Change in Conjunctival Hyperemia
Description: The change in proportion of participant's score will be analyzed. Rate of conjunctival hyperemia will be evaluated through the Efron scale which includes 5 grades: Normal (0), Very Mild (I), Mild (II), Moderate (3), and Severe (4). This outcome measure considered the Per Protocol (PP) population.
Time Frame: Days: 0 (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: In total, 18 participants were discontinued from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 46 | 49 | 40
Participants
  Elegibility visit: Normal | 21 | 15 | 14
  Elegibility visit: Very Mild | 14 | 17 | 12
  Elegibility visit: Mild | 9 | 15 | 11
  Elegibility visit: Moderate | 2 | 2 | 3
  Elegibility visit: Severe | 0 | 0 | 0
  First follow-up visit: Normal | 23 | 22 | 22
  First follow-up visit: Very Mild | 17 | 22 | 14
  First follow-up visit: Mild | 6 | 5 | 4
  First follow-up visit: Moderate | 0 | 0 | 0
  First follow-up visit: Severe | 0 | 0 | 0
  Final visit: Normal | 32 | 33 | 27
  Final visit: Very Mild | 11 | 14 | 13
  Final visit: Mild | 3 | 2 | 0
  Final visit: Moderate | 0 | 0 | 0
  Final visit: Severe | 0 | 0 | 0

6. Secondary Outcome: Incidence of Related Non Expected Adverse Events
Description: Number of related non expected adverse events observed per group. This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.
Time Frame: Days: 0 (eligibility visit), 0 - 2 (baseline visit),17 - 19 (± 1) (first follow-up visit), 31 - 33 (± 1) (final visit), and 38 - 40 (± 1) (safety call).
Measure: Number; unit: adverse events
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 61 | 61 | 60
adverse events | 5 | 5 | 10

7. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: With the patient's best possible refractive correction, visual acuity will be evaluated through the Snellen chart. Its notation (decimal) is described as the distance from the chart at which the test is performed, divided by the distance at which a letter equals vertically 5 minutes of arc.
  Visual acuity (VA) is a test of visual function. It will be evaluated with the Snellen chart. The Snellen chart is the standard tool used to evaluate visual acuity. It was located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20
Time Frame: Days: 0 (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Population: This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.
Measure: Mean (Standard Deviation); unit: decimal
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 61 | 61 | 60
decimal
  Elegibility visit | 0.97 (0.18) | 0.95 (0.21) | 0.94 (0.20)
  First follow-up visit | 0.99 (0.17) | 0.98 (0.26) | 0.96 (0.22)
  Final visit | 0.99 (0.2) | 0.96 (0.18) | 0.96 (0.22)

8. Secondary Outcome: Change in Incidence of Chemosis
Description: Chemosis will be evaluated as present (if conjunctiva separates from the sclera in ≥ 1/3 of the palpebral opening area or if it exceeds the eyelid's gray line) or absent per subject. This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.
Time Frame: Days: 0 (eligibility visit), 17 - 19 (± 1) (first follow-up visit), and 31 - 33 (± 1) (final visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
Number analyzed (Participants) | 61 | 61 | 60
Participants
  Elegibility visit | 0 | 0 | 0
  First follow-up visit | 0 | 0 | 0
  Final visit | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was recollected starting from the elegibility visit (day 0) until the security call (day 38 - 40) done at the end of the study. In this study, AE were collected during of 1 year, 5 months
Arm/Group | Arm 1; Humylub Ofteno® PF | Arm 2; Hyabak® | Arm 3; Lagricel Ofteno® PF
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 40/61 | 39/61 | 43/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1; Humylub Ofteno® PF (N=61) | Arm 2; Hyabak® (N=61) | Arm 3; Lagricel Ofteno® PF (N=60)
Convulsive Crisis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1; Humylub Ofteno® PF (N=61) | Arm 2; Hyabak® (N=61) | Arm 3; Lagricel Ofteno® PF (N=60)
Ocular burning (Eye disorders) | 27 (27) | 29 (33) | 30 (31)
Pruritus (Eye disorders) | 11 (12) | 5 (5) | 15 (15)
Ocular hyperemia (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 | 0 (0) | 3 (3)
Foreign body sensation in the eye (Eye disorders) | 5 (5) | 2 (2) | 9 (9)
Eyestrain (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Tearing (Eye disorders) | 2 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04702776/Prot_SAP_000.pdf